CLINICAL TRIAL: NCT03680092
Title: A Randomized Phase II Trial Comparing a Calcineurin Inhibitor-free Graft-versus-host Disease Prophylaxis Regimen With Post-transplantation Cyclophosphamide and Abatacept to Standard of Care
Brief Title: Comparing Cyclophosphamide and Abatacept With Standard of Care Treatment Following Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dimitrios Tzachanis, MD PhD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Dimitrios Tzachanis, MD PhD, Assistant Clinical Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180383
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: GVHD; Hematologic Neoplasms
Keywords: cancer; Graft-Versus-Host Disease; Hematologic Neoplasms; Abatacept; Cyclophosphamide; GVHD prophylaxis; stem cell transplantation; High risk hematologic malignancy; hematologic malignancy; Allogeneic Hematopoetic Stem Cell Transplantation; GVHD
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Graft vs Host Disease | interventions — Cyclophosphamide; Abatacept; Methotrexate; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide and abatacept (Experimental): The GVHD prophylaxis regimen on the experimental arm will consist of high dose Cyclophosphamide on Days +3 and +4 followed by abatacept for 6 months. Abatacept at a dose of 10mg/kg will be administered on days +5, +14 and +28, +56, +84, +112, +140, +168
  Interventions: Drug: Cyclophosphamide; Drug: abatacept
- methotrexate and tacrolimus (Active Comparator): The GVHD prophylaxis regimen on the standard of care arm will consist of methotrexate on Days +1,+3, +6 and +11 and tacrolimus
  Interventions: Drug: Methotrexate; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Day 3 and day 4 following transplant. Dosing will be based on patients' actual weight up to 120% of ideal body weight, above which it will be based on adjusted ideal body weight (ideal weight plus 50% of the difference between ideal and actual weight).
  Other Names: cytophosphane; Cytoxan; Neosar
  Arms: Cyclophosphamide and abatacept
Drug: abatacept — Abatacept at a dose of 10mg/kg will be administered on days +5, +14 and +28, +56, +84, +112, +140, +168
  Other Names: ORENCIA
  Arms: Cyclophosphamide and abatacept
Drug: Methotrexate — standard of care Methotrexate 5 mg/m2 on Days 1, 3, 6 and 11
  Other Names: Trexall
  Arms: methotrexate and tacrolimus
Drug: Tacrolimus — Tacrolimus per institutional guidelines
  Other Names: Prograf; Astagraf XL; Envarsus XR
  Arms: methotrexate and tacrolimus

SUMMARY:
The purpose of this study is to investigate whether the combination of cyclophosphamide and abatacept versus the treatment used in standard of care will reduce the incidence of moderate and severe chronic graft-versus-host disease (GVHD) following hematopoietic stem cell transplantation. GVHD occurs when the cells from your donor (the graft) see your body's cells (the host) as different and attack them.

DETAILED DESCRIPTION:
The experimental GVHD prophylaxis arm consists of cyclophosphamide and abatacept. Cyclophosphamide induces apoptosis of activated T cells and abatacept (CTLA4Ig) blocks activation of T cells by inhibiting the co-stimulatory signal.

Compared to the standard-of-care control arm, the experimental arm is much more convenient and expected to be associated with fewer toxicities.

In addition there is a great theoretical potential for immunological synergy between cyclophosphamide and abatacept for inducing post-transplant immunologic tolerance that clinically might translate into less GVHD without increase in relapse Patients will be randomized 1:1 to the experimental vs the standard of care arm. Randomization will be done prior to the use of any conditional therapy.

The two arms will be stratified by disease (acute leukemia vs others) and donor type (MRD vs MUD/MUD vs Haplo) in an effort to keep them balanced.

The conditioning regimen for both arms will be mainly Busulfan/Fludarabine (A Total Body Irradiation based conditioning regimen will be allowed for diseases such as ALL)

The GVHD prophylaxis regimen on the experimental arm will consist of high dose Cyclophosphamide on Days +3 and +4 followed by abatacept for 6 months.

The GVHD prophylaxis regimen on the standard of care arm will consist of methotrexate on Days +1,+3, +6 and +11 and tacrolimus for patients with a 10/10 matched related or unrelated donor and of high dose cyclophosphamide on Days +3 and +4 followed by tacrolimus and mycophenolate for patients with a haploidentical donor.

ELIGIBILITY:
Inclusion Criteria:

* High risk hematologic malignancy justifying the need for an allogeneic hematopoetic stem cell transplantation: AML, ALL, CML in accelerated or blast phase, MDS/MPN, NHL, Hodgkin lymphoma, and multiple myeloma
* Creatinine clearance > 40
* Adequate hepatic function
* Normal cardiac function (EF > 50%)

Exclusion Criteria:

* Patients with hematologic malignancies for which transplant is not the only curative option, such as AML with good or intermediate cytogenetics or molecular markers in CR1 or CML in chronic phase
* Inability to identify an 10/10 HLA-Matched Donor (related or unrelated) or a haploidentical donor
* Active malignant disease relapse
* Active, uncontrolled infection, uncontrolled cardiac angina, symptomatic congestive heart failure
* Life expectancy <3 months
* Pregnancy or lactation
* Patients may not be receiving any other investigational agents in the last 28 days
* Patients with chronic myeloid leukemia in first chronic phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tzachanis, MD PhD, Principal Investigator — University of California, San Diego; Divya Koura, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koura D, Dykes K, Goodman A, Costello C, Mulroney C, Mangan JK, Tanaka TN, Ball ED, Hamdan A, Jeong AR, Mirocha J, Zhang Q, Ogrodnik P, McConnell K, Maroge JJ, Padilla M, Morris GP, Tzachanis D. A prospective clinical trial of GVHD prophylaxis with posttransplant cyclophosphamide and abatacept. Blood Adv. 2025 Aug 26;9(16):4336-4344. doi: 10.1182/bloodadvances.2024015094. PMID 40554429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclophosphamide and Abatacept | Methotrexate and Tacrolimus
Started | 28 | 15
Completed | 25 | 15
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclophosphamide and Abatacept | Methotrexate and Tacrolimus | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 13 | 34
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 8 | 23
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Moderate and Severe Chronic GVHD at One Year Post Transplant
Description: The occurrence of moderate and severe chronic GVHD at one year post Chronic GVHD will be diagnosed and staged according to the previously published and widely accepted National Institutes of Health consensus criteria
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide and Abatacept | Methotrexate and Tacrolimus
Number analyzed (Participants) | 24 | 14
Participants | 0 | 8

2. Secondary Outcome: GVHD- and Relapse- Free Survival by One Year Post Transplant
Description: GVHD- and relapse- free survival will be defined as the absence of acute GVHD Grade III or IV or moderate or severe chronic GVHD or relapse or non-relapse mortality by one year post transplant. Acute GVHD will be diagnosed and graded according to Glucksberg criteria
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide and Abatacept | Methotrexate and Tacrolimus
Number analyzed (Participants) | 24 | 14
Participants | 15 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cyclophosphamide and Abatacept | Methotrexate and Tacrolimus
All-Cause Mortality (participants affected / at risk) | 2/25 | 3/15
Serious Adverse Events (participants affected / at risk) | 9/25 | 13/15
Other Adverse Events (participants affected / at risk) | 5/25 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide and Abatacept (N=25) | Methotrexate and Tacrolimus (N=15)
Febrile Neutropenia (Infections and infestations) | 4 (5) | 10 (11)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
CMV viremia (Infections and infestations) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (5)
Oral mucositis (Gastrointestinal disorders) | 2 (3) | 2 (3)
pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 6 (10) | 7 (11)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
hemorrhagic cystitis (Renal and urinary disorders) | 1 (1) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
C diff infection (Infections and infestations) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
engraftment syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
HLH (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hyperbilirubinemiα (Hepatobiliary disorders) | 0 (0) | 1 (5)
hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
hypogammaglobulinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hypokalemia (Renal and urinary disorders) | 0 (0) | 1 (2)
ischemic colitis and perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
PTLD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
retinal detachment (Eye disorders) | 0 (0) | 1 (1)
volume overload (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide and Abatacept (N=25) | Methotrexate and Tacrolimus (N=15)
CMV Viremia (Infections and infestations) | 5 (5) | 4 (6)
oral mucositis (Gastrointestinal disorders) | 3 (8) | 9 (13)
dry eyes (Eye disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 6 (9)
BK viremia (Infections and infestations) | 0 (0) | 2 (2)
colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
fatigue (General disorders) | 0 (0) | 5 (5)
fever (Infections and infestations) | 0 (0) | 3 (3)
EBV viremia (Immune system disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 0 (0) | 2 (3)
nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
TTP (Blood and lymphatic system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03680092/Prot_SAP_000.pdf